CLINICAL TRIAL: NCT02768207
Title: A Single Arm, Open Label, Phase II, Multicenter Study to Assess The Detection of The BRAF V600 Mutation on cfDNA From Plasma in Patients With Advanced Melanoma
Brief Title: A Study to Detect V-Raf Murine Sarcoma Viral Oncogene Homolog B1 (BRAF) V600 Mutation on Cell-Free Deoxyribonucleic Acid (cfDNA) From Plasma in Participants With Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ML29741; 2015-001731-20 (EudraCT Number)
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — cobimetinib; Vemurafenib

ARMS (1):
- Treatment Phase: Vemurafenib+Cobimetinib (Experimental): Participants with BRAF V600 mutation will receive vemurafenib 960 milligrams (mg) tablets orally twice daily (BID) on Days 1 to 28 along with cobimetinib 60 mg tablets orally once daily (OD) for 21 consecutive days (Days 1 to 21) of each 28-day cycle until disease progression, consent withdrawal, or the development of unacceptable toxicity.
  Interventions: Drug: Cobimetinib; Drug: Vemurafenib

INTERVENTIONS:
Drug: Cobimetinib — Participants will receive cobimetinib 60 mg tablets (three 20 mg tablet) orally OD for 21 consecutive days (Days 1 to 21), followed by a 7 day break (Days 22 to 28); in each 28-day cycle of treatment phase until disease progression, consent withdrawal, or the development of unacceptable toxicity.
  Other Names: GDC-0973, RO5514041, XL518
Drug: Vemurafenib — Participants will receive vemurafenib 960 mg tablets (four 240 mg tablet) orally BID from Day 1 to Day 28 of each 28-day cycle of the treatment phase until disease progression, consent withdrawal, or the development of unacceptable toxicity.
  Other Names: RO5185426

SUMMARY:
This is a single arm, multicenter, open label, and non-randomized clinical study on adult participants with unresectable or metastatic melanoma. The study will be conducted in two phases. Pre-screening phase will assess the BRAF V600 mutation in a new mutation analysis triggered by a mutant plasma cfDNA test result. Treatment phase will assess the clinical outcome for the participants treated with vemurafenib plus cobimetinib. The length of the study will be approximately 38 months.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening phase:

* Participants with histologically confirmed cutaneous melanoma, either unresectable Stage IIIc or Stage IV metastatic melanoma, as defined by American Joint Committee on Cancer 7th edition
* Documentation of BRAF V600 test result mutation-positive status on melanoma tumor tissue using a validated tissue test

Treatment Phase:

* Eastern Cooperative Oncology Group performance status of 0-2
* Adequate hematologic and end organ function obtained within 14 days prior to first dose of study drug treatment
* Negative serum pregnancy test prior to commencement of dosing in women of childbearing potential
* Absence of any psychological, familial, sociological, or geographical condition that potentially hampers compliance with the study protocol and treatment regimen and follow-up after treatment discontinuation schedule
* Female participants of childbearing potential and male participants with partners of childbearing potential must agree to always use two effective forms of contraception during the course of this study and for at least 6 months after completion of study therapy
* Participants should be able to swallow tablets
* Documentation of BRAF mutation positive status in melanoma tissue

Exclusion Criteria:

Treatment Phase:

* History of prior rapidly accelerated fibrosarcoma or mitogen-activated protein kinase pathway inhibitor treatment
* Use of prior chemotherapy or immunotherapy (including treatment with an anti-programmed death 1, or anti- programmed death ligand 1 or anti-cytotoxic T-lymphocyte-associated protein 4 monoclonal antibody) within 4 weeks before first study drug administration
* Palliative radiotherapy within 14 days prior to the first dose of study treatment
* Evidence of retinal pathology on ophthalmologic examination
* Systemic risk factors for retinal vein occlusion
* History of clinically significant cardiac dysfunction
* Current severe, uncontrolled systemic disease
* Pregnancy, lactating or breast feeding
* Intake of St. John's wort or hyperforin (a potent cytochrome P450 3A4 [CYP3A4 enzyme inducer] and grapefruit juice (a potent CYP3A4 enzyme inhibitor) at least 7 days prior to initiation of and during the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with BRAF V600 Mutation as Assessed Using the Idylla^TM Diagnostic Platform | Days -56 to -1 (Pre-screening period)
Concentration of BRAF V600 Mutation as Determined on Plasma cfDNA | Days -56 to -1 (Pre-screening period)
Number of Participants by BRAF Mutation Status | Days -56 to -1 (Pre-screening period)
Number of Participants with BRAF V600 Mutation as Assessed Using the Idylla^TM Diagnostic Platform in Participants With BRAF Wild-Type Based on a Prior Tissue Test Result | Days -56 to -1 (Pre-screening period)

SECONDARY OUTCOMES:
Percentage of Participants with Objective Response as Assessed by the Investigator According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Baseline up to disease progression or death whichever occurs first (up to 38 months)
Progression-Free Survival (PFS) | Baseline up to disease progression or death whichever occurs first (up to 38 months)
Duration of Response as Assessed by Investigator According to RECIST v1.1 | Baseline up to disease progression or death whichever occurs first (Up to 38 months)
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 Cycle 1 up to 4 weeks after end of treatment or until initiation of another anti-cancer therapy, whichever occurs first (up to 38 months)
Overall Survival | Baseline up to death (up to 38 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Belgium (11):
  - Institut Jules Bordet, Brussels
  - UZ Brussel, Brussels
  - CHIREC Edith Cavell, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - AZ Groeninge, Kortrijk
  - Clinique Ste-Elisabeth, Namur
  - AZ Delta (Campus Wilgenstraat), Roeselare
  - AZ Nikolaas (Sint Niklaas), Sint-Niklaas
  - Sint Augustinus Wilrijk, Wilrijk
- Poland (3):
  - Klinika Onkologii Klinicznej CO-I Kraków, Krakow
  - Szpital Kliniczny im. Heliodora Święcickiego UM w Poznaniu., Poznan
  - Centrum Onkologii- Instytut; im. M.Skłodowskiej-Curie, Warsaw